CLINICAL TRIAL: NCT05374681
Title: LEADH: Efficacy of a Minimally Invasive Therapy Adjuvant to the Standards of Care by Cyanoacrylate Embolization : Liquid Embolic Agent for the Treatment of Chronic subDural Hematoma a Randomized Control Study
Brief Title: Efficacy of a Minimally Invasive Therapy Adjuvant to the Standards of Care by Cyanoacrylate Embolization
Acronym: LEADH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29BRC22.0028
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Subdural Hematoma
Keywords: Cyanoacrylate; Embolization; Middle meningeal artery; Recurrence of chronic subdural hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Medical treatment alone (Other): Medical treatment without embolization of the MMA.
  Interventions: Other: Medical treatment
- Surgical treatment alone (Other): Surgical treatment without embolization of the MMA.
  Interventions: Other: Surgical treatment
- Medical treatment associated with an embolization of the MMA (Experimental): Medical treatment + embolization under local anesthesia or conscious sedation. The embolization will be carried out by femoral or radial arterial guided by pre-embolization cervical CTA. The middle meningeal artery will be catheterized then embolized by cyanoacrylates until the occlusion of the MMA.
  Interventions: Other: Medical treatment; Other: embolization of the MMA
- Surgical treatment associated with an embolization of the MMA (Experimental): Surgical treatment + embolization under local anesthesia or conscious sedation. The embolization will be carried out by femoral or radial arterial guided by pre-embolization cervical CTA. The middle meningeal artery will be catheterized then embolized by cyanoacrylates until the occlusion of the MMA.
  Interventions: Other: Surgical treatment; Other: embolization of the MMA

INTERVENTIONS:
Other: Medical treatment — Medical treatment alone
  Arms: Medical treatment alone; Medical treatment associated with an embolization of the MMA
Other: Surgical treatment — Surgical treatment alone
  Arms: Surgical treatment alone; Surgical treatment associated with an embolization of the MMA
Other: embolization of the MMA — The middle meningeal artery will be catheterized then embolized by cyanoacrylates until the occlusion of the MMA.
  Arms: Medical treatment associated with an embolization of the MMA; Surgical treatment associated with an embolization of the MMA

SUMMARY:
Chronic subdural hematomas (CSH) are collections of blood in the subdural space. CSH are becoming the most common cranial neurosurgical condition among adults, and a significant public health problem, due to an increasing use of anticoagulant and antiplatelet medication in an ageing population. Symptomatic CSH, or CSH with a significant mass effect, are treated surgically. However, recurrences are common (10 to 20%). Conservative management (medical) is used in patients who are asymptomatic or have minor symptoms. However, therapeutic failures, requiring surgical treatment, are common. The pathophysiology of CSH involves inflammation, angiogenesis, and clotting dysfunction. Self-perpetuation and rebleeding is thought to be caused by neo-membranes from the inflammatory remodeling of the dura-mater mainly fed by the distal branches of the middle meningeal artery (MMA). There are 13 ongoing registered RCTs in CSH, with the most common covering application of steroids, surgical techniques and tranexamic acid. Further to this, there are trials running on other pharmacological agents, and peri-operative management. Some industrial or academic trials are or will enroll in France in the next year in France. But to our best knowledge, none of these trials will the eventual benefits of the MMA embolization in both cases of medical and/or surgical management, and none will focus on the use of cyanoacrylates (CYA) for this purpose.

Preliminary case series and nonrandomized retrospective studies have suggested that MMA embolization alone or as adjuvant therapy to surgery can decrease recurrences.

The investigators hypothesize that in both conditions of conservative or surgical managements, endovascular embolization of patients with CSH significantly reduces the risk of recurrence of CSH. The investigators choose the CYA as liquid embolic agent because of the pain and cost of the use of Ethylen Vinyl alcohol copolymer (EVOH) agents and its simplicity to be used.

DETAILED DESCRIPTION:
* Indication of surgical or conservative management will be decided by the neurosurgeon.
* Experimental arm:

CSH requiring hematoma removal will be surgically managed with a surgical technique applied depending on the surgeon's discretion.

Medical management will be adopted according to neurosurgeons habits. MMA embolization (on the CSH side or bilaterally if necessary) in the Experimental Arms will be performed with Cyanoacrylates and preferentially using conscious sedation or local anesthesia.

• Control arm: CSH requiring hematoma removal will be surgically managed with a surgical technique applied depending on the surgeon's discretion.

Medical management will be adopted according to neurosurgeons habits

• Primary and secondary end points will be assessed at 2 months+/- 1 month and assessed at 6 +/- 2 months. The blind items will be the mRS and the RACE score. The volume of the CSH will be semi-automatically assessed using the ABC/2 method and the estimated maximal thickness of the CSH on axial images.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a more than 10 mm CSH confirmed by NCCT
* CSH localized to convexity
* Patient aged 18 years or more at the time of the enrollment
* Patient beneficiary from health insurance

Exclusion Criteria:

* Any contraindication as required per angiogram procedure (severe renal failure ≥ 4, allergy…)
* Pre-existing severe disability resulting in baseline mRS score > 3
* Life expectancy of less than 6 months due to another cause than CSH
* Patient under legal protection or deprived of liberty by a judicial or administrative decision
* Pregnant or breastfeeding women
* Vulnerable persons unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-09-28 (Estimated); Study Completion 2028-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of CSH recurrence defined by the composite endpoint | At 6 month
  CSH recurrence defined by the composite endpoint:
  * A symptomatic CSH during the 6 month FU period
  * A secondary surgical management during the 6 months FU period
  * A remaining or reaccumulated hematoma on NCCT at 6 months

SECONDARY OUTCOMES:
Number of symptomatic CSH during the FU period | At 6 month
  Number of symptomatic CSH during the FU period
Number of secondary surgical management during the FU period | At 6 month
  Number of secondary surgical management during the FU period
Number of remaining or reaccumulated hematoma on NCCT | At 6 month
  Number of remaining or reaccumulated hematoma on NCCT
Clinical efficacy | At 6 month
  Mortality rate
Clinical efficacy | At 6 month
  Shift Modified Rankin Scale (mRS) (min = 0 = better outcome, max = 5 = worse outcome)
Clinical efficacy | At 6 month
  Rapid Arterial oCclusion Exam (RACE) score evaluation (min = 0 = better outcome, max = 9 = worse outcome)
Clinical efficacy | At 6 month
  Quality of life of patients will be evaluated by the EuroQol-5Dimensions-5L questionnaire
Clinical efficacy | At 6 month
  Neurological exam : Barthel Scale (min = 0 = worse outcome, max = 100 = better outcome)
Success rate of the embolization (success = technical success of the procedure. Failure of the procedure = total or partial (catheterization, injection, other)). | At 6 month
  Success rate of the embolization (success = technical success of the procedure. Failure of the procedure = total or partial (catheterization, injection, other)).
Complication rate of the embolization | At 6 month
  Complication rate of the embolization
Volumetry of the CSH, calculated by the ABC/2 method. | At 6 month
  Volumetry of the CSH, calculated by the ABC/2 method.
Maximum thickness of the CSH in mm. | At 6 month
  Maximum thickness of the CSH in mm.
Comparison of the rate of AE in both groups | At 6 month
  Comparison of the rate of AE in both groups
Comparison of the rate of SAE in both groups | At 6 month
  Comparison of the rate of SAE in both groups

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU Amiens-Picardie, Amiens, France
  - CHU Brest, Brest, France
  - CHU Caen, Caen, France
  - Hôpital Henri Mondor, Créteil, France
  - CHU Nantes, Nantes, France
  - CHU Nice, Nice, France
  - Hôpital Pitié Salpêtrière, Paris, France
  - Hôpital Fondation Rothschild, Paris, France
  - CHU Tours, Tours, France
  - CHU Bordeaux, Bordeaux
  - CHU Nancy, Nancy

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.